CLINICAL TRIAL: NCT02657369
Title: An Open-Label, Single-Arm, Multicenter, Phase 2 Trial of Lenvatinib for the Treatment of Anaplastic Thyroid Cancer (ATC)
Brief Title: A Phase 2 Trial of Lenvatinib for the Treatment of Anaplastic Thyroid Cancer (ATC)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Overall response rate was 3% (only 1 out of 33 participants had confirmed PR).
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E7080-M000-213; 2015-001929-17 (EudraCT Number)
Record Dates: First submitted 2016-01-13; First posted 2016-01-15 (Estimated); Results first posted 2019-10-15 (Actual); Last update posted 2019-10-15 (Actual); Status verified 2017-11

CONDITIONS: Thyroid Carcinoma, Anaplastic
Keywords: Lenvatinib; Thyroid Cancer, Anaplastic; Lenvima; E7080
MeSH Terms: conditions — Thyroid Carcinoma, Anaplastic | interventions — lenvatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes

ARMS (1):
- Lenvatinib (Experimental): Participants will receive lenvatinib 24 milligrams (mg) (2 10-mg capsules and one 4-mg capsule) once daily by oral administration at approximately the same time each morning for up to approximately 24 months.
  Interventions: Drug: Lenvatinib 24 mg

INTERVENTIONS:
Drug: Lenvatinib 24 mg
  Other Names: Lenvima; E7080

SUMMARY:
The primary purpose of the study is to evaluate objective response rate ([ORR]: complete response [CR] and partial response [PR]) by investigator review in participants with anaplastic thyroid cancer (ATC) treated with lenvatinib.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must have histological diagnosis consistent of Anaplastic Thyroid Cancer (ATC). Cytologic diagnosis by fine needle aspiration alone is not sufficient. Histologic diagnosis may be made by core needle biopsy, incisional biopsy, thyroidectomy, or other surgical biopsy. Fresh tumor biopsies (re-biopsy) should be obtained whenever feasible. The central pathology review may take place prior to or after the participant starts treatment with lenvatinib.

   1. Central review of pathology is required for study participation, but not required prior to enrollment or start of treatment in order to avoid delay. If the results of central pathology review are not available prior to the start of study treatment, the confirmation of diagnosis of ATC at the local laboratory is mandatory prior to scheduled start of treatment with lenvatinib.
   2. If central pathology review indicates a diagnosis other than ATC, the participant may continue treatment with lenvatinib per standard of care, at the discretion of the treating investigator. Participants deemed to have another diagnosis (not ATC) will be taken off this study and replaced for the purpose of efficacy analyses.
   3. Differentiated thyroid carcinoma (DTC) with focus loci of ATC is allowed. If a participant has pathology showing a small focus of ATC arising out of DTC and the measurable disease is not fully consistent with ATC, confirmation of ATC by biopsy is required.
   4. An incidental focus of medullary thyroid cancer (MTC), DTC, and/or poorly differentiated thyroid cancer in a participant with ATC is allowed.
   5. Histological diagnosis of ATC made through surgical resection is also acceptable.
2. Prior neoadjuvant, adjuvant, or palliative chemotherapy for ATC is allowed.
3. Measurable disease based on investigator's assessments meeting the following criteria:

   1. At least 1 lesion of ≥ 10 millimeters (mm) in the longest diameter for a non-lymph node or ≥ 15 mm in the short-axis diameter for a lymph node which is serially measurable according to Response Evaluation Criteria In Solid Tumors (RECIST) 1.1 using computerized tomography (CT) or magnetic resonance imaging (MRI).
   2. Lesions that have had external beam radiotherapy or locoregional therapies such as radiofrequency ablation must show evidence of subsequent progressive disease (substantial size increase of ≥ 20%) to be deemed a target lesion.
4. Participants with known brain metastases who have completed whole brain radiotherapy, stereotactic radiosurgery, or complete surgical resection will be eligible if they have remained clinically stable, asymptomatic, and off steroids for 1 month prior to enrollment.
5. All previous chemotherapy or radiation therapy-related toxicities, except dry mouth, dysphagia, esophagitis, mucositis, alopecia, and irreversible late sequelae of radiation therapy, must have resolved to Grade 0 or 1 per Common Terminology Criteria for Adverse Events (CTCAE v 4.03), and all wounds from prior surgery must have adequately recovered.
6. Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1.
7. Blood pressure (BP) ≤ 140/90 millimeter of mercury (mmHg) at screening with or without antihypertensive medications and no change in antihypertensive medications within 1 week prior to Cycle 1/Day 1.
8. Adequate renal function as evidenced by calculated creatinine clearance ≥ 30 milliliter/ minute (mL/min) according to the Cockcroft and Gault formula.
9. Adequate bone marrow function:

   1. Absolute neutrophil count (ANC) ≥ 1.5 x 10^9/liter (L) and
   2. Hemoglobin ≥ 9.0 grams/deciliter (g/dL) (can be corrected by growth factor or transfusion) and
   3. Platelet count ≥ 100 x 10^9/L.
10. Adequate blood coagulation function as evidenced by an International Normalized Ratio (INR) ≤ 1.5.
11. Adequate liver function:

    1. Bilirubin ≤ 1.5 x upper limit of normal (ULN) except for unconjugated hyperbilirubinemia or Gilbert's syndrome;
    2. Alkaline phosphatase (ALP), alanine aminotransferase (ALT), and aspartate aminotransferase (AST) ≤ 3 x ULN (≤ 5 x ULN if participant has liver metastases). If ALP is > 3 x ULN (in the absence of liver metastases) or > 5 x ULN (in the presence of liver metastases) AND participants are also known to have bone metastases, the liver-specific ALP must be separated from the total and used to assess the liver function instead of the total ALP.
12. Voluntary agreement to provide written informed consent and the willingness and ability to comply with all aspects of the protocol.

Exclusion Criteria:

1. Differentiated thyroid cancer (DTC) or MTC. However, ATC arising out of DTC is allowed, as long as the measurable disease is clinically consistent with ATC i.e., rapidly progressive and/or 18F fluorodeoxyglucose (FDG)-avid.
2. Newly diagnosed participants who are considered appropriate candidates for comprehensive multimodality treatment (involving surgery and/or external beam radiotherapy or chemo radiotherapy).
3. Prior treatment with lenvatinib or any tyrosine kinase inhibitor (TKI) - (except for combination therapy of radiation and reduced dose of TKI given for the purpose of radiosensitization).
4. Major surgery within 2 weeks prior to the first dose of lenvatinib.
5. Any anti-cancer treatment within 14 days or any investigational agent within 30 days before the first dose of study drug.
6. Radiotherapy within 3 weeks prior to the first dose of lenvatinib.
7. Participants having > 1 + proteinuria on urine dipstick testing will undergo 24 hour urine collection for quantitative assessment of proteinuria. Participants with urine protein ≥ 1 gram/24 hours will be ineligible.
8. Significant cardiovascular impairment: History of (a) congestive heart failure greater than New York Heart Association (NYHA) Class II, (b) unstable angina, (c) myocardial infarction, (d) stroke, or (e) cardiac arrhythmia associated with impairment within 6 months of the first dose of study drug.
9. A clinically significant electrocardiogram (ECG) abnormality, including a marked Baseline prolonged QT/QTc interval (e.g., a repeated demonstration of a QTc interval >500 milliseconds (msec)).
10. Active infection requiring systemic therapy.
11. Clinically significant hemoptysis or tumor bleeding within two weeks prior to first dose of lenvatinib.
12. Radiographic evidence of major blood vessel invasion/infiltration.
13. Other active malignancy (except definitively treated melanoma in-situ, basal or squamous cell carcinoma of the skin, or carcinoma in-situ of the cervix or bladder) within past 24 months.
14. Scheduled for major surgery during the study.
15. Females who are breastfeeding or pregnant at Screening or Baseline (as documented by a positive beta-human chorionic gonadotropin [ß-hCG] or human chorionic gonadotropin [hCG] test with a minimum sensitivity of 25 international units/liter (IU/L) or equivalent units of ß-hCG [or hCG]). A separate Baseline assessment is required if a negative screening pregnancy test was obtained more than 72 hours before the first dose of study drug.
16. Females of childbearing potential who:

    1. Do not agree to use a highly effective method of contraception (ie, total abstinence, [if it is their preferred and usual lifestyle], an intrauterine device or intrauterine system, a contraceptive implant, an oral contraceptive, or have a vasectomized partner with confirmed azoospermia) within 30 days before study entry and throughout the entire study period and for 30 days after study drug discontinuation.
    2. Are currently totally abstinent (as their preferred and usual lifestyle), and who do not agree to be totally abstinent during the study period and for 30 days after study drug discontinuation.
    3. Are using hormonal contraceptives but are not on a stable dose of the same hormonal contraceptive product for at least 4 weeks before dosing and who do not agree to use the same contraceptive during the study and for 30 days after study drug discontinuation.
    4. Are using oral hormonal contraceptives and who do not agree to add a barrier method.

    (NOTE: All females will be considered to be of childbearing potential unless they are postmenopausal [amenorrheic for at least 12 consecutive months, in the appropriate age group, and without other known or suspected cause] or have been sterilized surgically [i.e. bilateral tubal ligation, total hysterectomy, or bilateral oophorectomy, all with surgery at least 1 month before dosing]).

    For sites outside of the European Union (EU), it is permissible that if a highly effective method of contraception is not appropriate or acceptable to the subject, then the subject must agree to use a medically acceptable method of contraception, i.e. double barrier methods of contraception such as condom plus diaphragm or cervical/vault cap with spermicide.
17. Evidence of clinically significant disease (e.g., cardiovascular, respiratory, gastrointestinal, renal disease) that in the opinion of the investigator(s) could affect the participant's safety or interfere with the study assessments.
18. Known intolerance to the study drug or any of the excipients.
19. Any medical or other condition that in the opinion of the investigator(s) would preclude the participant's participation in a clinical study.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2016-07-07 (Actual); Primary Completion 2018-09-26 (Actual); Study Completion 2018-09-26 (Actual)

CONTACTS AND LOCATIONS:
Locations (26):
- United States (12):
  - Scottsdale, Arizona
  - Duarte, California
  - Washington D.C., District of Columbia
  - Jacksonville, Florida
  - Miami, Florida
  - Boston, Massachusetts
  - Rochester, Minnesota
  - New York, New York
  - Durham, North Carolina
  - Portland, Oregon
  - Philadelphia, Pennsylvania
  - Houston, Texas
- Australia (2):
  - Camperdown, New South Wales
  - St Leonards, New South Wales
- France (5):
  - Caen, Calvados
  - Bordeaux, Gironde
  - Angers, Maine Et Loire
  - Lyon, Rhone
  - Villejuif, Val De Marne
- Italy (4):
  - Milan
  - Pisa
  - Roma
  - Siena
- United Kingdom (3):
  - Cardiff, South Glamorgan
  - Glasgow, Strathclyde
  - Sutton, Surrey

IPD SHARING:
Plan to Share IPD: Yes
Eisai IPD sharing statement: Eisai's data sharing commitment and further information on how to request data can be found on our website http://eisaiclinicaltrials.com/.

REFERENCES:
- [Derived] Wirth LJ, Brose MS, Sherman EJ, Licitra L, Schlumberger M, Sherman SI, Bible KC, Robinson B, Rodien P, Godbert Y, De La Fouchardiere C, Newbold K, Nutting C, Misir S, Xie R, Almonte A, Ye W, Cabanillas ME. Open-Label, Single-Arm, Multicenter, Phase II Trial of Lenvatinib for the Treatment of Patients With Anaplastic Thyroid Cancer. J Clin Oncol. 2021 Jul 20;39(21):2359-2366. doi: 10.1200/JCO.20.03093. Epub 2021 May 7. PMID 33961488
- [Derived] Cabanillas ME, McFadden DG, Durante C. Thyroid cancer. Lancet. 2016 Dec 3;388(10061):2783-2795. doi: 10.1016/S0140-6736(16)30172-6. Epub 2016 May 27. PMID 27240885

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 13 investigative sites in France, Italy, United Kingdom, Australia and the United States from 07 July 2016 to 26 September 2018.
Pre-assignment Details: A total of 48 participants were screened, of which 14 were screen failures and 34 were enrolled to receive study treatment.
Groups:
- Lenvatinib 24 mg: Participants received lenvatinib 24 milligram (mg) (two 10-mg capsules and one 4-mg capsule), orally, once daily in a 28-days treatment cycle up to disease progression, development of unacceptable toxicity, lost to follow up, withdrawal of consent, participant's choice, pregnancy, or study termination by sponsor (approximately 27 months).
Period: Overall Study
Arm/Group | Lenvatinib 24 mg
Started | 34
Completed | 0
Not Completed | 34
Not completed — Death | 27
Not completed — Study terminated by sponsor | 7

BASELINE CHARACTERISTICS:
Population: The full analysis set included all participants who received at least one dose of lenvatinib.
Groups:
- Lenvatinib 24 mg: Participants received lenvatinib 24 mg (two 10-mg capsules and one 4-mg capsule), orally, once daily in a 28-days treatment cycle up to disease progression, development of unacceptable toxicity, lost to follow up, withdrawal of consent, participant's choice, pregnancy, or study termination by sponsor (approximately 27 months).
Arm/Group | Lenvatinib 24 mg
Number analyzed (Participants) | 34
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.4 (10.09)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 29
  Unknown or Not Reported | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 27
  More than one race | 0
  Unknown or Not Reported | 3

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR)
Description: ORR was defined as the percentage of participants with best overall response (BOR) of complete response (CR) or partial response (PR) as determined by investigator review using Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 for target lesions. CR was defined as disappearance of all target lesions. All pathological lymph nodes (whether target or non-target) must have a reduction in their short axis to less than 10 millimeter (mm). PR was defined as at least a 30 percent (%) decrease in the sum of the longest diameters of target lesions, taking as reference the Baseline sum diameters. Confirmation of CR or PR was performed at least 28 days following the initial achievement of the response.
Time Frame: From the date of beginning of lenvatinib administration to the date of first documentation of disease progression or death, whichever occurred first (up to Month 27)
Population: The evaluable analysis set included all participants with histological diagnosis of ATC that was confirmed by central pathology review and who received at least one dose of lenvatinib.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Lenvatinib 24 mg
Number analyzed (Participants) | 33
percentage of participants | 3.0 [0.1 to 15.8]

2. Secondary Outcome: Progression-free Survival (PFS) Rate
Description: Twelve-week PFS rate was the percentage of participants in the analysis population who remain alive and progression-free at 12 weeks. PFS was defined as the time from the date of beginning of lenvatinib administration to the date of first documentation of confirmed disease progression or death, whichever occurred first. The Kaplan-Meier estimated rate method was used to estimate 12-week PFS, along with the corresponding 95% confidence interval (CI). Participants who were off study due to lost to follow up, withdrew consent, or study terminated by sponsor, had new anti-cancer treatment, had no baseline/post-baseline tumor assessments, or missed 2 or more visits prior to event were censored.
Time Frame: From the date of beginning of lenvatinib administration up to the date of first documentation of confirmed disease progression or death, whichever occurred first (up to Week 12)
Population: The full analysis set included all participants who received at least one dose of lenvatinib.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Lenvatinib 24 mg
Number analyzed (Participants) | 34
percentage of participants | 36.4 [20.6 to 52.3]

3. Secondary Outcome: Overall Survival (OS) Rate
Description: Six-month OS rate was defined as the percentage of participants in the analysis population who are alive at 6 months. OS was defined as the time from the date of beginning of lenvatinib administration until date of death from any cause. The Kaplan-Meier estimated rate method was used to estimate six-month OS, along with the corresponding 95% CI. Participants with last known alive date as study terminated by sponsor were censored.
Time Frame: From the date of beginning of lenvatinib administration up to date of death from any cause (up to Month 6)
Population: The full analysis set included all participants who received at least one dose of lenvatinib.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Lenvatinib 24 mg
Number analyzed (Participants) | 34
percentage of participants | 41.2 [24.8 to 56.9]

4. Secondary Outcome: Median PFS
Description: PFS was defined as the time from the date of beginning of lenvatinib administration to the date of first documentation of confirmed disease progression or death, whichever occurs first. Median PFS was estimated using the Kaplan-Meier method. Participants who were off study due to lost to follow up, withdrew consent, or study terminated by sponsor, had new anti-cancer treatment, had no baseline/post-baseline tumor assessments, or missed 2 or more visits prior to event were censored.
Time Frame: From the date of beginning of lenvatinib administration to the date of first documentation of confirmed disease progression or death, whichever occurred first (up to Month 27)
Population: The full analysis set included all participants who received at least one dose of lenvatinib.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Lenvatinib 24 mg
Number analyzed (Participants) | 34
months | 2.6 [1.4 to 2.8]

5. Secondary Outcome: Median OS
Description: OS was defined as the time from the date of beginning of lenvatinib administration until date of death from any cause. Median OS was estimated using the Kaplan-Meier method. Participants with last known alive date as study terminated by sponsor were censored.
Time Frame: From the date of beginning of lenvatinib administration up to date of death from any cause (up to Month 27)
Population: The full analysis set included all participants who received at least one dose of lenvatinib.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Lenvatinib 24 mg
Number analyzed (Participants) | 34
months | 3.2 [2.8 to 8.2]

ADVERSE EVENTS:
Time Frame: From signature of informed consent form up to 28 days after last dose of study drug (up to Month 27)
Groups:
- Lenvatinib: Participants received lenvatinib 24 mg (two 10-mg capsules and one 4-mg capsule), orally, once daily in a 28-days treatment cycle up to disease progression, development of unacceptable toxicity, lost to follow up, withdrawal of consent, participant's choice, pregnancy, or study termination by sponsor (approximately 27 months).
Arm/Group | Lenvatinib
All-Cause Mortality (participants affected / at risk) | 27/34
Serious Adverse Events (participants affected / at risk) | 25/34
Other Adverse Events (participants affected / at risk) | 32/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lenvatinib (N=34)
Deep vein thrombosis (Vascular disorders) | 1 (1)
Hypertension (Vascular disorders) | 2 (2)
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 10 (10)
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Metastases to peritoneum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Asthenia (General disorders) | 2 (2)
Chest pain (General disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1)
Pyrexia (General disorders) | 2 (2)
Confusional state (Psychiatric disorders) | 1 (1)
Accidental overdose (Injury, poisoning and procedural complications) | 1 (1)
Cardiopulmonary failure (Cardiac disorders) | 1 (2)
Abdominal lymphadenopathy (Blood and lymphatic system disorders) | 1 (1)
Agranulocytosis (Blood and lymphatic system disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Tracheal fistula (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Presyncope (Nervous system disorders) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Anal fistula (Gastrointestinal disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 2 (3)
Odynophagia (Gastrointestinal disorders) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (2)
Renal failure (Renal and urinary disorders) | 1 (2)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 2 (2)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (2)
Abscess neck (Infections and infestations) | 1 (1)
Anal abscess (Infections and infestations) | 1 (1)
Arthritis infective (Infections and infestations) | 1 (1)
Bacterial sepsis (Infections and infestations) | 1 (1)
Perirectal abscess (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Pyelitis (Infections and infestations) | 1 (1)
Septic shock (Infections and infestations) | 1 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lenvatinib (N=34)
Bloody discharge (Vascular disorders) | 1 (1)
Hypertension (Vascular disorders) | 18 (34)
Hypotension (Vascular disorders) | 2 (2)
Inferior vena cava dilatation (Vascular disorders) | 1 (1)
Vena cava thrombosis (Vascular disorders) | 1 (1)
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (3)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Contrast media reaction (Immune system disorders) | 1 (1)
Asthenia (General disorders) | 5 (8)
Cyst (General disorders) | 1 (1)
Facial pain (General disorders) | 1 (1)
Fatigue (General disorders) | 11 (14)
Injection site bruising (General disorders) | 1 (1)
Localised oedema (General disorders) | 1 (1)
Malaise (General disorders) | 2 (2)
Mucosal inflammation (General disorders) | 1 (1)
Oedema peripheral (General disorders) | 2 (2)
Pain (General disorders) | 2 (4)
Anxiety (Psychiatric disorders) | 2 (2)
Depressed mood (Psychiatric disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 3 (3)
Arthropod bite (Injury, poisoning and procedural complications) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Post procedural complication (Injury, poisoning and procedural complications) | 1 (1)
Post procedural swelling (Injury, poisoning and procedural complications) | 1 (1)
Postoperative delirium (Injury, poisoning and procedural complications) | 1 (1)
Stoma site pain (Injury, poisoning and procedural complications) | 1 (1)
Alanine aminotransferase increased (Investigations) | 2 (3)
Aspartate aminotransferase increased (Investigations) | 3 (3)
Bilirubin conjugated increased (Investigations) | 2 (2)
Blood alkaline phosphatase increased (Investigations) | 3 (4)
Blood bilirubin increased (Investigations) | 2 (2)
Blood creatinine increased (Investigations) | 1 (1)
Blood phosphorus increased (Investigations) | 1 (1)
Blood thyroid stimulating hormone decreased (Investigations) | 1 (1)
Blood thyroid stimulating hormone increased (Investigations) | 3 (3)
C-reactive protein increased (Investigations) | 1 (1)
Electrocardiogram QT prolonged (Investigations) | 2 (2)
Gamma-glutamyltransferase increased (Investigations) | 2 (4)
International normalised ratio increased (Investigations) | 3 (3)
Liver function test abnormal (Investigations) | 1 (1)
Lymphocyte count decreased (Investigations) | 4 (5)
Oxygen saturation decreased (Investigations) | 1 (1)
Platelet count decreased (Investigations) | 2 (2)
Sputum normal (Investigations) | 1 (1)
Troponin increased (Investigations) | 1 (1)
Urine analysis abnormal (Investigations) | 1 (2)
Urine leukocyte esterase positive (Investigations) | 1 (1)
Weight decreased (Investigations) | 9 (12)
White blood cell count decreased (Investigations) | 2 (2)
Acute myocardial infarction (Cardiac disorders) | 1 (1)
Atrial tachycardia (Cardiac disorders) | 1 (1)
Hyperdynamic left ventricle (Cardiac disorders) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 1 (1)
Bronchial secretion retention (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (5)
Dry throat (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 5 (8)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 (5)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 (5)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 6 (8)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Nasal obstruction (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 6 (10)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 2 (2)
Increased tendency to bruise (Blood and lymphatic system disorders) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1)
Lymphopenia (Blood and lymphatic system disorders) | 2 (3)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Amnesia (Nervous system disorders) | 1 (1)
Cervical radiculopathy (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 4 (4)
Dysgeusia (Nervous system disorders) | 3 (5)
Facial paralysis (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 5 (6)
Hyperaesthesia (Nervous system disorders) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 1 (1)
Jugular vein occlusion (Nervous system disorders) | 1 (1)
Lethargy (Nervous system disorders) | 1 (1)
Somnolence (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Tremor (Nervous system disorders) | 1 (1)
Vision blurred (Eye disorders) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 3 (3)
Vertigo (Ear and labyrinth disorders) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 3 (5)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 2 (3)
Anal fistula (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 7 (8)
Dental caries (Gastrointestinal disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 8 (13)
Diverticulum (Gastrointestinal disorders) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 3 (4)
Dyspepsia (Gastrointestinal disorders) | 3 (3)
Dysphagia (Gastrointestinal disorders) | 7 (10)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1)
Gingival pain (Gastrointestinal disorders) | 2 (4)
Gingival recession (Gastrointestinal disorders) | 1 (1)
Glossodynia (Gastrointestinal disorders) | 2 (6)
Haemorrhoids (Gastrointestinal disorders) | 1 (1)
Loose tooth (Gastrointestinal disorders) | 1 (1)
Mouth swelling (Gastrointestinal disorders) | 1 (1)
Mouth ulceration (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 11 (17)
Odynophagia (Gastrointestinal disorders) | 2 (3)
Oesophageal stenosis (Gastrointestinal disorders) | 1 (1)
Oral dysaesthesia (Gastrointestinal disorders) | 1 (1)
Oral mucosal erythema (Gastrointestinal disorders) | 1 (1)
Oral pain (Gastrointestinal disorders) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1)
Periodontal disease (Gastrointestinal disorders) | 1 (1)
Proctalgia (Gastrointestinal disorders) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 10 (13)
Tongue dry (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 6 (9)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1)
Proteinuria (Renal and urinary disorders) | 8 (15)
Pyelocaliectasis (Renal and urinary disorders) | 1 (2)
Cholecystitis (Hepatobiliary disorders) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1)
Cholestasis (Hepatobiliary disorders) | 1 (1)
Gallbladder enlargement (Hepatobiliary disorders) | 1 (2)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 2 (2)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 2 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 2 (2)
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 1 (1)
Macule (Skin and subcutaneous tissue disorders) | 1 (1)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 8 (9)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (3)
Pruritus generalised (Skin and subcutaneous tissue disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Rash macular (Skin and subcutaneous tissue disorders) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (3)
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 (1)
Skin discolouration (Skin and subcutaneous tissue disorders) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 (8)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (5)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Bursitis (Musculoskeletal and connective tissue disorders) | 1 (1)
Coccydynia (Musculoskeletal and connective tissue disorders) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 (2)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 4 (4)
Neck pain (Musculoskeletal and connective tissue disorders) | 4 (5)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Hypothyroidism (Endocrine disorders) | 6 (6)
Decreased appetite (Metabolism and nutrition disorders) | 10 (12)
Dehydration (Metabolism and nutrition disorders) | 2 (2)
Hypercalcaemia (Metabolism and nutrition disorders) | 3 (3)
Hyperglycaemia (Metabolism and nutrition disorders) | 5 (5)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1)
Hyperuricaemia (Metabolism and nutrition disorders) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2 (2)
Hypocalcaemia (Metabolism and nutrition disorders) | 2 (4)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 3 (3)
Hyponatraemia (Metabolism and nutrition disorders) | 9 (15)
Hypophagia (Metabolism and nutrition disorders) | 1 (1)
Arthritis infective (Infections and infestations) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1)
Oral candidiasis (Infections and infestations) | 3 (3)
Paronychia (Infections and infestations) | 1 (1)
Perirectal abscess (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Superinfection (Infections and infestations) | 1 (1)
Tooth infection (Infections and infestations) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 2 (2)
Urinary tract infection (Infections and infestations) | 4 (4)

LIMITATIONS AND CAVEATS:
The study was terminated since overall response rate was 3% (only 1 out of 33 participants had confirmed PR).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2016-05-24): https://cdn.clinicaltrials.gov/large-docs/69/NCT02657369/Prot_000.pdf
  • Statistical Analysis Plan (2018-10-18): https://cdn.clinicaltrials.gov/large-docs/69/NCT02657369/SAP_001.pdf